CLINICAL TRIAL: NCT05303181
Title: The Effect of Different Russian Current Parameters on Maximum Voluntary Isometric Contraction(MVIC) of the Quadriceps Muscle Among University of Sharjah Students: A Randomized Controlled Trail.
Brief Title: The Effect of Different Russian Current Parameters on MVIC Contraction of the Quadriceps Muscle Among University of Sharjah Students.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ansam Tayseer Hasan, principal investigator, University of Sharjah
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: REC-21-02-18-01-S
Record Dates: First submitted 2022-02-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (Experimental): training used Russian Current carrier frequency at 2500-Hz alternating current.
  Interventions: Device: Russian Current
- Group2 (Experimental): training used Russian Current carrier frequency at 3750-Hz alternating current.
  Interventions: Device: Russian Current
- Group3 (Experimental): training used Russian Current carrier frequency at 5000-Hz alternating current.
  Interventions: Device: Russian Current
- Group4 (Experimental): training used Russian Current at different mode.
  Interventions: Device: Russian Current

INTERVENTIONS:
Device: Russian Current — The patient will be placed in sitting position, hip at 90-degree flexion, knee at 60°, the upper body supported by the backrest, cross belt support the trunk and cross belt support the pelvis. The dynamometer rotating axis will be aligned with knee joint axis and the resistance lever arm will place in the distal leg above the malleolus. The angle of the joints adjustment considering the joint's range of motion and the device's user's manual, any movement other than the range of motion determined by the mechanical limit will be not allowed
  All electrical induced contraction will last 4 second each, with characteristics of 75 bursts; 4 second time on, 400 μs pulse width and 10 second time off. The greatest electrically induced torque by the quadriceps muscle at the maximum current output from the stimulator will be recorded for each subject to be used in data analysis. The same procedure will be done on the 3rd week and after 6th week.
  Other Names: The Biodex isokinetic dynamometer

SUMMARY:
The study aims to investigate the effect of different Russian current parameters on maximum voluntary isometric contraction of the quadriceps muscle among University of Sharjah students.

DETAILED DESCRIPTION:
Muscular strength and endurance are two important compatible parts of the body; for normal people to move, lift things and do day-to-day activities or athletic performance. Large number of studies have been carried out to elaborate the different factor that help in improving the muscular strength as well as the endurance combined with rehabilitation programs in order to promote muscle function and prevent the injury(Akinoglu & Kocahan, 2020; Chou & Binder-Macleod, 2007; Evetovich et al., 2001; Selkowitz, 1985; Snyder-Mackler et al., 1994; Ward et al., 2006). Strengthening and endurance training have been used frequently in varied rehabilitation protocols in order to improve the overall musculoskeletal performance.(Earl & Hoch, 2011; Gondin et al., 2011). Meanwhile, Isokinetic training and Neuromuscular electrical stimulation are frequently utilized in physical therapy.(Brown & Whitehurst, 2003; Chou & Binder-Macleod, 2007; Evetovich et al., 2001; Stone, 1997).

Russian current is one of the popular preferred Neuromuscular electrical stimulation as it has been advocated to increase muscle strength due to its high tolerance as well as minimum pain level provocation (Akinoglu & Kocahan, 2020; Gondin et al., 2011). Russian currents are alternating currents at a frequency of 2.5 kHz that are burst modulated at a frequency of 50 Hz with a 50% duty cycle. The widely and most popular training protocol used with Russian current is (10/50/10) in which the stimulus is applied for a 10-second "on" period followed by a 50-second "off" or rest period, with a recommended treatment time of 10 minutes per stimulation session. Russian currents are used mainly to generate a motor response, but it also has been investigated as an electro-analgesia type intervention. This training protocol is used mainly to generate a motor response, but it also has been investigated as an electro-analgesia type intervention.

Despite a lot of previous research regarding the Russian current; no studies are available in which suggest the most efficient carrier frequency for Russian current to strengthening the muscles and increase muscle with isokinetic training in the short term and the effect of different RC on the EIT by the quadriceps muscle. The aim of this study is directed toward investigation of those different Russian current carrier frequencies' effects on the quadriceps muscle isokinetic strength and endurance in addition to investigate the effect of different mode of RC on the EIT by the quadriceps femoris muscle. This study will include measurement for the knee torque and quadriceps muscle strength using Biodex system 3 that will be generated by different carrier frequency in addition to different RC mode, and investigate the relationship between those variables.

ELIGIBILITY:
Inclusion Criteria:

1. Their age ranged from 18 to 25 years.
2. Their Body Mass Index (BMI) within normal range (18.5-25).
3. Don't have any health related condition that required medical attention in the past two years.
4. All participant at same physical fitness level.

Exclusion Criteria:

* The subjects will be excluded from this study if they have any of the following criteria:

  1. Quadriceps muscle injury.
  2. Spinal or lower limb fractures.
  3. Lower limb deformities.
  4. Associated cognition abnormalities which may to affect muscle and limb function
  5. Tumors or radicular symptoms
  6. Recent muscular lesion, knee injury, sensory changes and neuromuscular disease
  7. Previous surgery that may affect the lower limb muscle performance.
  8. Any contraindication for Russian current application

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-08 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
establish the relationship between the different carrier frequency for burst modulated electrical stimulation as an independent variable and electrical induced quadriceps femoris muscle torque (EIT) as a dependent variable. | measured data will be recorded at the 3rd week after training using RC and at 6th week as a follow up measurements
  The primary outcome of the study is to establish the relationship between the different carrier frequency for burst modulated electrical stimulation as an independent variable and electrical induced quadriceps femoris muscle torque (EIT) as a dependent variable.
  And the effect of different RC mode on the electrical induce torque by the quadriceps muscle. The EIT measurement will be done using the Biodex pro 3 system devices this system was described in detail; with reliability and validity has been investigated previous study establish its reliable. This study, will investigate the effect of different carrier frequency 2500Hz-3750Hz-5000Hz alternating current on the electrical induce quadriceps muscle torque of the dominant leg, and the effect of different Russian current mode on the EIT of the quadriceps muscle femoris.

IPD SHARING:
Plan to Share IPD: No
All information taken will be kept confidential and will not be taken without the participant's consent. Any data collected will be for scientific purpose only.The therapists have been instructed about the privacy, confidentiality and rights of the participants .
  Published data will remain anonymous without personal identifier of participants